CLINICAL TRIAL: NCT05817032
Title: Effect of Telerehabilitation Practice in Long COVID-19 Patients: Impact on Stress Oxidative, Inflammation, Functional Capacity and Quality of Life
Brief Title: Effect of Telerehabilitation Practice in Long COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Nurul Paramita, dr, M.Biomed, SpKFR, Indonesia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-07-0713
Record Dates: First submitted 2023-04-16; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Long COVID-19; Long COVID; Post COVID-19 Condition; Post-COVID-19 Syndrome; Post-COVID Syndrome
Keywords: Long COVID-19; Telerehabilitation; rehabilitation; exercise
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Motor Activity | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Experimental): Baseline measurement will be done in the rehabilitation center. Prescription for rehabilitation will be determined based on the result of baseline measurement. Participants will receive rehabilitation intervention that include telerehabilitation (video conference regular meeting, text message reminder, and mobile app). Participants will attend a regular check up at the center once a month. After 12 weeks post intervention measurement will be taken.
  Interventions: Behavioral: Telerehabilitation
- Control group (Active Comparator): Baseline measurement will be done in the rehabilitation center. Prescription for rehabilitation will be determined based on the result of baseline measurement. Participants will be given instruction how to do proper exercise training at home. Participants will attend a regular check up at the center once a month. After 12 weeks post intervention measurement will be taken.
  Interventions: Behavioral: Standard rehabilitation care

INTERVENTIONS:
Behavioral: Telerehabilitation — Exercise prescriptions will be given based on the result of baseline assessment. The intensity of the exercise prescription and level of monitoring will be tailored to each participant's ability and condition. Exercise will be prescribed by a Physical Medicine and Rehabilitation specialist in accordance with standard rehabilitation protocols. Exercise will consist of aerobic exercise, resistance exercise and breathing exercise. Participants are asked to commit to do at least 36 sessions of exercise. Participants will be allowed to have a hybrid approach (10-12 in person, 24-26 virtual) or fully virtual.
  Arms: Telerehabilitation group
Behavioral: Standard rehabilitation care — Exercise prescriptions will be given based on the result of baseline assessment. The intensity of the exercise prescription and level of monitoring will be tailored to each participant's ability and condition. Exercise will be prescribed by a Physical Medicine and Rehabilitation specialist in accordance with standard rehabilitation protocols. Exercise will consist of aerobic exercise, resistance exercise and breathing exercise. Participants are asked to commit to do at least 36 sessions of exercise. Participants will be allowed to have 10-12 in person exercise.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to test the efficacy of telerehabilitation practice in Long COVID-19 patients. The main question[s] it aims to answer are whether telerehabilitation practice in Long COVID-19 patients help to reduce stress oxidative, reduce inflammation, improve functional capacity and improve quality of life.

Participants will receive 12 weeks of telerehabilitation practice Researchers will compare intervention group (that received telerehabilitation) and control group (that received standard treatment) to see if there is better outcome in intervention group.

DETAILED DESCRIPTION:
Study background:

Several study show that some survivors of COVID-19 have post COVID-19 sequelae. Previous studies suggest that rehabilitation interventions with appropriate prescription of physical exercise can provide short, medium and long term health benefits. Telerehabilitation services are an innovative strategy to support rehabilitation intervention and hopefully able to increase compliance of patients to exercise program.

This study aims to prove the effectiveness of telerehabilitation in improving levels of inflammation, oxidative stress, functional capacity and quality of life in Long COVID-19 patients. Participants will be divided into intervention group and control group. Baseline measurement will be taken. Telerehabilitation will be given to the intervention group for 12 weeks. Control group will receive standard rehabilitation treatment. After 12 weeks post intervention measurement will be taken.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 survivors
* Have at least one of the following sequelae:
* fatigue
* dyspnea and/or chronic cough
* joint and/or muscle pain
* headache
* insomnia (difficulty sleeping)
* impaired concentration / memory
* Willing to take part in the telerehabilitation program regularly during the study
* Willing to participate in the research and sign the consent form

Exclusion Criteria:

* Unable to use the mobile phone application and zoom meet
* Unable to come to the hospital for examination or training (if needed)
* Cognitive impairment (MMSE <21)
* Neuromusculoskeletal disorder which will affect rehabilitation interventions
* Severe chronic lung disease
* Severe heart disease (Grade III-IV from the New York Heart Association)
* Chronic kidney disorders
* Malignancy
* Severe autoimmune disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in quality of life status measured using European Quality of Life 5 Dimension 5 Level (EQ 5D 5L) questionnaire at 12 weeks | Baseline and week 12
  European Quality of Life 5 Dimension 5 Level (EQ 5D 5L) questionnaire is a validated instrument to measure quality of life. It is a descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Change from baseline the distance from Six Minute Walk Test at 12 weeks | Baseline and week 12
  Six minute walk test is a validated instrument developed by the American Thoracic Society and it was officially introduced in 2002, coming along with a comprehensive guideline. The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Change from baseline the mean Glutathione (GSH)/ oxidized GSH (GSSG) ratio at 12 weeks | Baseline and week 12
  The ratio of reduced Glutathione (GSH) to oxidized GSH (GSSG) is an indicator of cellular health, with reduced GSH constituting up to 98% of cellular GSH under normal conditions. It will be measured using The Glutathione GSH/GSSG Assay Kit, which is designed to accurately measure total, reduced and oxidized glutathione in biological samples using an enzymatic method that utilizes Ellman's Reagent (DTNB) and glutathione reductase (GR).
Change from baseline the mean endothelial microparticles at 12 weeks | Baseline and week 12
  Endothelial microparticles is an emerging marker of endothelial dysfunction and also considered to play a major biological role in inflammation, vascular injury, angiogenesis, and thrombosis. Techniques to measure circulating endothelial microparticles rely on differential centrifugation in platelet-free plasma and on the identification of cell-surface Cluster of Differentiations (CD) antigens.

SECONDARY OUTCOMES:
Change from baseline the score from Brief Fatigue Inventory (BFI) questionnaire at 12 weeks | Baseline and 12 weeks
  Brief Fatigue Inventory (BFI) questionnaire is a valid instrument to assess the severity of fatigue and the impact of fatigue on daily functioning. A global fatigue score can be obtained by averaging all the items on the BFI.
Change from baseline the score from hand grip strength test using handgrip dynamometer at 12 weeks | Baseline and 12 weeks
  The purpose of the handgrip strength test is to measure the maximum isometric strength of the hand and forearm muscles. Handgrip strength is important because people with strong hands tend to be strong elsewhere, so this test is often used as a general test of strength.

CONTACTS AND LOCATIONS:
Overall Officials: Nurul Paramita, MD, MBiomed, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Fakultas Kedokteran Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
individual participant data including study protocol and informed consent available upon personal request